CLINICAL TRIAL: NCT00021658
Title: Effects of Pesticide Exposure on Neurodevelopment/Growth/Respiratory Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Clinica de Salud (Other); Natividad Medical Center (Other)
Purpose: Prevention
Other Study IDs: 9605-CP-001
Record Dates: First submitted 2001-07-30; First posted 2001-08-01 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-07

CONDITIONS: Environmental Exposure
Keywords: Epidemiology; pesticide; asthma; children; exposure
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Procedure: Pesticide application procedures

SUMMARY:
Exposure and health study of pesticide and allergen exposures to pregnant women and children. Intervention study is planned after assessment is completed.

DETAILED DESCRIPTION:
Exposure assessment and pathway analysis of organophosphate pesticides to low income pregnant women and children living in the Salinas valley of California. Health study investigating neurodevelopment, growth, and asthma in children.

ELIGIBILITY:
* Female, at least 18 years of age.
* Live in Salinas valley in California.
* Pregnant.
* Medical eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550
Dates: Start 1999-10; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Eskenazi, Ph.D., Principal Investigator — University of California at Berkeley; Asa Bradman, Ph.D., Study Director — University of California at Berkeley
Locations (1):
- CHAMACOS Field Office, Salinas, California, United States